CLINICAL TRIAL: NCT06365164
Title: Presence of the Rooting Reflex on Preterms' ? Study of the Emergence of Sensory Self-awareness in Premature Newborns: Comparison of the Rooting Reflex Response Between Facilitated Self-stimulation and External Stimulation
Brief Title: Study of the Emergence of Sensory Self-awareness in Premature Newborns Using the Rooting Reflex
Acronym: PREMATACT
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Faculty of Psychology and Educational Sciences,University of Geneva (Unknown)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0354
Record Dates: First submitted 2024-03-21; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: Premature; Development, Child; Rooting Reflex
Keywords: rooting reflex; sensory self-awareness; tactile sensory; premature newborn; development care
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Premature newborns: Children born prematurely between 28 and 37 weeks of amenorrhoea, aged at least 3 days.
  Interventions: Behavioral: Tactile stimulation

INTERVENTIONS:
Behavioral: Tactile stimulation — The procedure consists of brief perioral tactile stimulation. The procedure is filmed in order to record and evaluate the response of the newborn to the stimulation. During the same intervention, each newborn will receive external stimulation (the experimenter repeatedly and regularly touches the corner of the infant's mouth slowly with the tip of his index finger) followed by facilitated self-stimulation (the experimenter will place the newborn's elbow close to his body, allowing him to touch his face alone with his hand). There will also be an initial phase and a final 30-second phase in which the newborn is observed without any stimulation.

SUMMARY:
The main objective is to demonstrate the presence of the rooting reflex in premature and the emergence of sensory self-awareness in premature by showing a difference in the response of the rooting reflex to external tactile stimulation and to facilitated tactile self-stimulation during quiet wakefulness.

The main hypothesis is to confirm the tactile skills of the very premature newborn in exploring the rooting reflex and then to evaluate the emergence of sensory self-awareness.

The investigators assume a difference in response in favour of a greater response of the newborn to external tactile stimulation compared to facilitated self-stimulation in favour of the distinction between self and non-self showing the emergence of a sensory awareness of self in the preterm newborn.

DETAILED DESCRIPTION:
Touch is the first sense to develop in foetal life. Children born prematurely have early tactile skills, in particular the ability to discriminate and learn. These tactile skills can be expressed through the newborn's reflexes. The sensory exploration that takes place when reflexes are manifested can be the basis for tactile learning and, in particular, for the development of the baby's awareness of his own body, with discrimination of the self. As touch plays an essential role in the child's perceptual-cognitive development, studying the tactile skills of premature infants is an ideal approach for a better understanding of the development of primitive sensory awareness.

The main hypothesis is to confirm the tactile skills of the very premature newborn in exploring the rooting reflex and then to evaluate the emergence of sensory self-awareness, by comparing the response of the rooting reflex between facilitated self-stimulation and external stimulation.

The investigators assume a difference in response in favour of a greater response of the newborn to external tactile stimulation compared to facilitated self-stimulation in favour of the distinction between self and non-self showing the emergence of a sensory awareness of self in the preterm newborn.

The study of the specific sensory of the premature newborn is part of the continuum of developmental care, and is part of an approach to improving the care delivered in neonatology with the aim of encouraging the best neurological development.

ELIGIBILITY:
Inclusion Criteria:

* Children born prematurely between 28 and 37 weeks of amenorrhoea, aged at least 3 days.

Exclusion Criteria: Premature newborns with :

* respiratory assistance (invasive or non-invasive ventilation)
* malformative syndrome
* a genetic syndrome
* neurological damage such as stage III or IV intraventricular haemorrhage or periventricular leukomalacia,
* sedative treatment: morphine, clonidine
* aminergic treatment
* acute pathology: shock, sepsis, acute cardiac failure, acute respiratory failure, etc.

Ages: 28 Weeks to 37 Weeks | Sex: All
Age Groups: Child
Study Population: Children born prematurely between 28 and 37 weeks of amenorrhoea, aged at least 3 days.
Sampling Method: Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The emergence of sensory self-awareness in premature newborns by showing a difference in the response of the rooting reflex to external tactile stimulation and to facilitated tactile self-stimulation during calm awakening. | The data will be collected for one year. Each newborn baby can be included for 14 weeks.The intervention is 5 to 10 minutes corresponding to external stimulation and facilitated self-stimulation spaced at least 2 hours apart and for up to 48 hours.
  First the external stimulation procedure is 30-second phase of observation. Next, the experimenter touches the corner of the infant's mouth and repeatedly with his index finger (about 5 gentle touches of about 10 seconds, repeated about 5 times) depending on the state and commitment of the newborn, ending with a final observation period of 30 seconds.
  The facilitated self-stimulation procedure will begin and end with a 30-second observation period. Then the experimenter will place the newborn's elbow close to his body, allowing him to touch his face alone with his hand, on one side then the other, for 30 seconds, with 2 to 5 trials depending on the child's level of commitment.
  The coding use a qualitative scale of four behaviours from 1 to 4 that are increasingly representative of the rooting reflex. The primary outcome is defined by an average score of the relative frequencies representative of the rooting reflex and will be compared between the two stimulation conditions.

SECONDARY OUTCOMES:
The secondary objective is to show a longitudinal progression in the emergence of the rooting reflex by repeated inclusions (seven days minimum) at different terms for the same newborn. | Each subject will be able to take part in up to three interventions, each at least 7 days apart, until they reach 41 weeks' gestation. The data will be collected for one year. Each newborn baby can be included for 14 weeks.
  After inclusion, each subject will be able to take part in up to three interventions, each at least 7 days apart, until they reach 41 weeks' gestation.The investigators will use a qualitative scale of four behaviours from 1 to 4 that are increasingly representative of the rooting reflex :
  1. outward movement of the head
  2. movement of the head towards the stimulation
  3. movement of the head towards facial stimulation with the mouth open
  4. head movement towards facial stimulation with tongue protrusion. The fourth behaviour corresponds to the most complete rooting reflex, and is the highest score.
  For each newborn, the relative frequency of each of the four behaviours described above as gradually representative of the expression of the rooting reflex in the same newborn will be compared at different terms and according to the type of stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Doutau, Principal Investigator — University Grenoble Hospital
Locations (1):
- University Hospital Grenoble, Grenoble, Isere, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lejeune F, Marcus L, Berne-Audeoud F, Streri A, Debillon T, Gentaz E. Intermanual transfer of shapes in preterm human infants from 33 to 34 + 6 weeks postconceptional age. Child Dev. 2012 May-Jun;83(3):794-800. doi: 10.1111/j.1467-8624.2012.01753.x. Epub 2012 Mar 30. PMID 22469180
- [Background] Marcus L, Lejeune F, Berne-Audeoud F, Gentaz E, Debillon T. Tactile sensory capacity of the preterm infant: manual perception of shape from 28 gestational weeks. Pediatrics. 2012 Jul;130(1):e88-94. doi: 10.1542/peds.2011-3357. Epub 2012 Jun 25. PMID 22732168
- [Background] Als H, McAnulty GB. The Newborn Individualized Developmental Care and Assessment Program (NIDCAP) with Kangaroo Mother Care (KMC): Comprehensive Care for Preterm Infants. Curr Womens Health Rev. 2011 Aug;7(3):288-301. doi: 10.2174/157340411796355216. PMID 25473384
- See also: Study of Rochat about rooting reflex and sensory awareness in newborns — https://psychology.emory.edu/cognition/rochat/lab/DifferentialRootingResponse.pdf
- See also: Touch in premature newborns — https://scholar.archive.org/work/hsnqb7adbbdf5mqrdfjfusr7zi/access/wayback/https://www.cairn.info/load_pdf.php?ID_ARTICLE=ENF1_131_0033&download=1